CLINICAL TRIAL: NCT06440603
Title: Erythroid Krüppel Like Factor (EKLF) Gene Expression in β-thalassemia Patients
Brief Title: EKLF Gene Expression in β-thalassemia
Status: Not yet recruiting | Type: Observational
Sponsor: Rofaida Hassan Ahmed (Other)
Responsible Party: Sponsor-Investigator, Rofaida Hassan Ahmed, Principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: β-thalassemia
Record Dates: First submitted 2024-05-19; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: β-thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Ethylenediamine tetra-acetic acid (EDTA) peripheral blood samples 3- Reverse transcription-quantitative polymerase chain reaction (RT-qPCR) for detection of EKLF:
  * The method of total RNA extraction: TRIZOL and TRIZOL LS.
  * The purity and concentration of the RNA will be measured using Nano Drop 2000 instument.
  * cDNA will be done with primers using thr Goscript Reverse Transcription System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: Age and sex matched healthy Control
  Interventions: Diagnostic Test: PCR
- Group 2: 50 patients with β-thalassemia major
  Interventions: Diagnostic Test: PCR
- Group 3: 50 patients with β-thalassemia intermedia
  Interventions: Diagnostic Test: PCR

INTERVENTIONS:
Diagnostic Test: PCR — Reverse transcription-quantitative polymerase chain reaction (RT-qPCR) for detection of EKLF:
  * The method of total RNA extraction: TRIZOL and TRIZOL LS.
  * The purity and concentration of the RNA will be measured using Nano Drop 2000 instument.
  * cDNA will be done with primers using thr Goscript Reverse Transcription System

SUMMARY:
1. Studying the effect of expression pattern of EKLF gene in β-thalassemic patients.
2. Detecting the correlation between the gene expression of EKLF and the clinical phenotype of β-thalassemic patients.

DETAILED DESCRIPTION:
β-thalassemia is a common inherited disorder caused by absent or reduced synthesis of the hemoglobin subunit beta (beta globin chain) , it has 3 clinical types; minor which is a carrier state, intermedia and major which are differentiated by blood transfusion dependency and lab findings.

In β-thalassemia, insufficient production of the β-globin molecule results in an excess of free α-globin chains that can precipitate within erythroid precursors, impairing their maturation and leads to death of these precursors and ineffective production of erythroid cells. As a result, a significant anaemia occurs and the consequent expansion of erythroid precursors can lead to secondary problems in bones and other organs.

These mutations are primarily point mutations that affect transcriptional control, translation, and splicing of the beta haemoglobin gene and gene expression.

The frequency of beta-thalassemia mutations varies by regions of the world with the highest prevalence in the Mediterranean, the Middle East, and Southeast and Central Asia. Approximately 68000 children are born with beta-thalassemia. Its prevalence is 80-90 million carriers, around 1.5% of the global population.

Erythroid Krüppel-like factor (EKLF or KLF1) is a transcriptional regulator that plays a major role in lineage-restricted control of gene expression. KLF1 expression and activity are tightly controlled in a temporal and differentiation stage-specific manner. The mechanisms by which KLF1 is regulated encompass a range of biological processes, including control of KLF1 RNA transcription, protein stability, localization, and posttranslational modifications. Intact KLF1 regulation is essential to correctly regulate erythroid function by gene transcription and to maintain hematopoietic lineage homeostasis by ensuring a proper balance of erythroid/megakaryocytic differentiation. In turn, KLF1 regulates erythroid biology by a wide variety of mechanisms, including gene activation and repression by regulation of chromatin configuration, transcriptional initiation and elongation, and localization of gene loci to transcription factories in the nucleus.

Previous studies have shown that EKLF plays a critical role in regulating the developmental switch between fetal and adult haemoglobin expression, both by direct activation of β-globin and indirect repression of γ-globin gene expression in adult erythroid progenitors via regulation of Bcl11a and ZBTB7a and PUM1.

PUM1 is a direct posttranscriptional regulator of β-globin switching, whose expression is regulated by the erythroid master transcription factor erythroid Krüppel-like factor (EKLF/KLF1), peaks during erythroid differentiation, binds γ-globin messenger RNA (mRNA), and reduces γ-globin (HBG1) mRNA stability and translational efficiency, which culminates in reduced γ-globin protein levels.

So, EKLF is too important in erythropoiesis and Hb switching that there are clinical trials nowadays depending on the molecules that targeted by EKLF (eg:Bcl11a, ZBTB7a and PUM1) and their role in Hb switching in treatment of thalassemia and other haemolytic anaemias as sickle cell anaemia.

ELIGIBILITY:
Inclusion Criteria:

* patients with β-thalassemia (major and intermedia).
* patients are of both sexes (male or female) at any age

Exclusion Criteria:

* patients with any other types of hemolytic anaemia

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients > 5 years diagnosed with β-thalassemia including both thalassemia major and intermedia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
study the expression pattern of EKLF gene in β-thalassemic patients, work by measuring mRNA levels | Baseline
  study the expression pattern of EKLF gene by Real-time polymerase chain reaction (RT-qPCR) in β-thalassemic patients

SECONDARY OUTCOMES:
study the correlation between the gene expression of EKLF and the clinical phenotype of β-thalassemic patients. | Baseline
  study the correlation between the gene expression of EKLF and the clinical phenotype of β-thalassemic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Naser Eldin, Study Director — Assiut University; Sherif Helmy, Study Director — Assiut University; Reem Elagoz, Study Director — Assiut University

REFERENCES:
- [Background] Sankaran VG, Orkin SH. The switch from fetal to adult hemoglobin. Cold Spring Harb Perspect Med. 2013 Jan 1;3(1):a011643. doi: 10.1101/cshperspect.a011643. PMID 23209159
- [Background] Cao A, Galanello R. Beta-thalassemia. Genet Med. 2010 Feb;12(2):61-76. doi: 10.1097/GIM.0b013e3181cd68ed. PMID 20098328
- [Background] Origa R. beta-Thalassemia. Genet Med. 2017 Jun;19(6):609-619. doi: 10.1038/gim.2016.173. Epub 2016 Nov 3. PMID 27811859
- [Background] Yien YY, Bieker JJ. EKLF/KLF1, a tissue-restricted integrator of transcriptional control, chromatin remodeling, and lineage determination. Mol Cell Biol. 2013 Jan;33(1):4-13. doi: 10.1128/MCB.01058-12. Epub 2012 Oct 22. PMID 23090966
- [Background] Borg J, Papadopoulos P, Georgitsi M, Gutierrez L, Grech G, Fanis P, Phylactides M, Verkerk AJ, van der Spek PJ, Scerri CA, Cassar W, Galdies R, van Ijcken W, Ozgur Z, Gillemans N, Hou J, Bugeja M, Grosveld FG, von Lindern M, Felice AE, Patrinos GP, Philipsen S. Haploinsufficiency for the erythroid transcription factor KLF1 causes hereditary persistence of fetal hemoglobin. Nat Genet. 2010 Sep;42(9):801-5. doi: 10.1038/ng.630. Epub 2010 Aug 1. PMID 20676099
- [Background] Elagooz R, Dhara AR, Gott RM, Adams SE, White RA, Ghosh A, Ganguly S, Man Y, Owusu-Ansah A, Mian OY, Gurkan UA, Komar AA, Ramamoorthy M, Gnanapragasam MN. PUM1 mediates the posttranscriptional regulation of human fetal hemoglobin. Blood Adv. 2022 Dec 13;6(23):6016-6022. doi: 10.1182/bloodadvances.2021006730. PMID 35667093
- [Background] Siatecka M, Soni S, Planutis A, Bieker JJ. Transcriptional activity of erythroid Kruppel-like factor (EKLF/KLF1) modulated by PIAS3 (protein inhibitor of activated STAT3). J Biol Chem. 2015 Apr 10;290(15):9929-40. doi: 10.1074/jbc.M114.610246. Epub 2015 Feb 24. PMID 25713074